CLINICAL TRIAL: NCT05011435
Title: Assessment of the Feasibility of Using a Smartphone Application for the Prevention and Screening of Burnout
Brief Title: Assessment of the Feasibility of Using a Smartphone Application for the Prevention and Screening of Burnout (BURNOUT ADVICE)
Acronym: BURNOUT ADVICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weprom (Other)
Collaborators: Kelindi (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-2021-01
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-08

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users: users of the web-application
  Interventions: Device: web-application for burnout

INTERVENTIONS:
Device: web-application for burnout — Use of burnout advisor web-application for detection of professional burnout
  Other Names: Burnout Advisor

SUMMARY:
Burnout syndrome has been recognized as a mental illness since 2020. All workers can be affected. The consequences are multiple and often serious, ranging from stoppage of work to depression or even suicide. According to a 2019 survey by Malakoff, 56% of employees are in "professional or personal fragility", but the statistics are incomplete.

In the medical community, the burnout rate is doubled compared to the general population.

The diagnosis of pre-burnout can precede a burnout by several months, an early treatment can then reduce complications and improve the quality of life at work.

On a study model on health data already carried out as part of a cancer detection application in smokers which involved 7000 users and which showed the ability to of such an application to detect curable symptomatic cancers from questionnaires (24% with application against 9% without application), we will carry out a descriptive evaluation of the use of an application to detect pre-burnout, burnout and depressive syndrome in a worker population. In the event of a risk alert of pre-burnout, burnout or depressive syndrome, the application will display a message to the user suggesting that he consult his general practitioner or put him in contact with a doctor through a teleconsultation via a dedicated platform.

This first study will assess the feasibility and acceptability of an early detection approach among professionals of a state of "fragility" (pre-burnout, burnout or depressive syndrome). Subsequently, a larger study will evaluate the effectiveness of this application for the early detection of burnout among professionals, its management and the reduction of costs for the healthcare system and society.

ELIGIBILITY:
Inclusion Criteria:

* Person aged 18 to 64
* Exercising a professional activity
* User informed of the use of this data and not objecting to it

Exclusion Criteria:

* Professionals on sick leave

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population will include the first 200 users of the application who did not object to the use of their data for this assessment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
usefulness | 6 months
  number of users who find the application useful

SECONDARY OUTCOMES:
alert | 6 months
  Description of alerts triggered by algorithms
Consultation | 6 months
  Number of relevant consultations (or teleconsultations) after an alert

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, Pr, Study Director — ILC
Locations (1):
- ILC, Le Mans, France

IPD SHARING:
Plan to Share IPD: No